CLINICAL TRIAL: NCT04934358
Title: Effectiveness of a Follow-up Program Based on Motivational Interventions and Physical Exercise in Patients With Fragility Fracture: Randomized Controlled Clinical Trial.
Brief Title: Motivational Interventions and Physical Exercise in Patients With Fragility Fracture
Acronym: PREVFRAILTY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIGE-0040-2020
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Fragility Fracture
Keywords: fragility fracture; physical exercise; motivational intervention
MeSH Terms: conditions — Motor Activity | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity program and motivational intervention (Experimental): Physical activity program agreed with the patient / family and according to functional status (based on the 6-minute walk test) and motivational intervention. In addition to the care provided in usual care, a progressive physical exercise program based on basal functional capacity is prescribed. The exercise will be developed at home.
  Interventions: Behavioral: Physical and motivational follow-up treatment
- Treatment as usual (Active Comparator): Multidisciplinary rehabilitation provided by professionals in the hospital and primary care settings, according to the individual needs of patients at different times of their recovery and the accessibility and availability of services in the different care settings.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Physical and motivational follow-up treatment — Physical and motivational follow-up treatment
  Arms: Physical activity program and motivational intervention
Behavioral: Usual care — Usual rehabilitation program
  Arms: Treatment as usual

SUMMARY:
Patients with a fragility fracture are twice as likely to have future fractures compared to their non-fractured peers. Furthermore, the 30% who suffer a fragility fracture do not regain the level of functioning in terms of activities of daily living after one year. A recent ecological study, in several European countries, estimates that if fracture patients were enrolled in fracture follow-up services, at least 19,000 fractures could be prevented each year. Clinical trials carried out in the research group have shown that the prescription of physical exercise in severe underlying pathologies is effective in improving physical function, quality of life and long-term results.

Hypothesis: The implementation of a motivational intervention and physical exercise program, in a staggered manner, taking into account the basic exercise capacity, improves the functional status of the patient (basic activities of daily life), adherence to interventions and the level of physical activity, and therefore reduces the number of hospital admissions, refractures and other associated complications.

Objective: To evaluate the effect of a rehabilitation intervention based on physical exercise and motivation, applied in a staggered manner and according to the functional capacity of patients with fragility fracture.

DETAILED DESCRIPTION:
Method: Single-blind, randomized, controlled clinical study, with 2 parallel arms and single-center. Study subjects: Patients who underwent surgery for a fragility hip fracture between September 2021 and September 2022 in a tertiary hospital in southern Spain. A progressive physical exercise and motivational intervention adjusted for functional capacity will be compared versus usual rehabilitation care. Follow-up of patients for 3 months and a final visit at 6 months. The primary outcome variables will be functional status for the development of activities of daily living (individual ability to care for himself) and number of hospital readmissions (reasons and consequences). Variables related to quality of life, cognitive status, laboratory markers and densitometry will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Present a hip fracture (includes cervical fracture and trochanteric), classified in the 10th version of the International Classification of Diseases (ICD-10-ES) with codes S72-S72.26X;
* In addition, the fracture must be due to fragility: fracture due to a low-energy trauma or not proportional to the consequences (Hermoso de Mendoza, 2003);
* To have received a surgical repair by replacement arthroplasty or internal fixation (ICD-10-ES procedures: 0SU and 0SR) in a period of less than one week;
* To be recovering in a trauma and orthopedic unit and/or be transferred to a rehabilitation unit or discharged;
* Before the fracture, independent or mild dependence for activities of daily living (Barthel index> 60) and living at home;
* To have the cognitive ability to give informed consent (ANNEX I);
* To live and be domiciled in a basic health area covered by the study hospital complex
* To be over 50 years of age

Exclusion Criteria:

* Presence of low cognitive level (scores below 23 points in Lobo's Mini-cognitive exam);
* Patients with pathological fractures due to skeletal alterations other than osteoporosis;
* Presence of more than one fall (other than the cause of hospital admission) in the last year;
* Presence of uncorrected anemia (hemoglobin concentration <9/dL), acute infectious disease (C-reactive protein> 10 mg / L), severe cardiorespiratory disease (for example: unstable angina; severe heart failure identified by the New York Heart Association as class III-IV), musculoskeletal or neurological diseases (for example, major amputation of lower limbs) that make physical exercise impossible.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Barthel index | 6 months
  Functional status for the development of activities of daily living (individual ability to take care of himself)
Number of hospital readmissions | 6 months
  Other clinical outcomes, such as mortality and all-cause hospitalization,

SECONDARY OUTCOMES:
Mini-Mental State Examination | 6 months
  A 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment
Minnesota Leisure Time Physical Activity Questionnaire | 6 months
  To assess the quantity (total activity metabolic index) and quality (heavy, moderate, and light) of physical activity performed
Geriatric Depression Scale | 6 months
  is a brief, 30-item questionnaire in which participants are asked to respond by answering yes or no in reference to how they felt over the past week
Visual analogue scale | 6 months
  A validated, subjective measure for acute and chronic pain
Falls Efficacy Scale-International | 6 months
  It is a 16 item questionnaire, useful to the researchers and clinicians interested in fear of falling, with a score ranging from minimum 16 (no concern about falling) to maximum 64 (severe concern about falling)
5-level EQ-5D version | 6 months
  A standardised measure of health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Maimónides Biomedical Research Institute of Córdoba, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Segura-Ruiz R, Ruiz-Canete M, Munoz-Alonso A, Rivas-Cruces C, Serrano-Lazaro P, Armenteros-Ortiz PJ, Hidalgo-Lopezosa P, Lamberti N, Manfredini F, Lopez-Soto PJ. Effectiveness of a home-based physical exercise intervention in patients with fragility fractures on functional independence and hospital readmissions: a protocol for a randomised controlled trial. BMJ Open. 2025 Nov 4;15(11):e101342. doi: 10.1136/bmjopen-2025-101342. PMID 41248369